CLINICAL TRIAL: NCT05764694
Title: Correlation Between Occurrence of Bullying, Victimization and Deleterious Oral Habits Among School Children in Cairo Governorate, Egypt: Cross-Sectional Study
Brief Title: Correlation Between the Occurrence of School Bullying, Victimization, and the Occurrence of Deleterious Oral Habits.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yousra el-sayed taha, General dentist at the Egyptian Ministry of Health, Cairo University
Other Study IDs: effect of bullying on children
Record Dates: First submitted 2023-02-28; First posted 2023-03-13 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Bruxism; Nail Biting; Bullying of Child; Bullying
MeSH Terms: conditions — Bruxism; Nail Biting; Bullying

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: bullied children — A questionnaire will be answered by parent to measure the primary outcome of the study, which is Presence, duration, and frequency of Oral habits (Bruxism, Nail biting) in addition to a questionnaire answered by child to measure the secondary outcome which is Prevalence of Bullying and victimization.

SUMMARY:
To determine the correlation between the occurrence of bullying, victimization, and deleterious oral habit in a group of Egyptian school children.

DETAILED DESCRIPTION:
Bullying is a major educational and public health problem among school-aged children that has a short and long negative effect on their physiological and psychosocial health.

Bullying among school children is widely spreading and has different forms including physical as hitting, kicking, or verbal as an insult social as spreading rumors or the social exclusion or psychological as stalking or cyberbullying as online hacking.

Bullying affects children greatly in different manners as lack of self-esteem, lack of concentration, depression, anxiety, and expressing feeling of loneliness. The World Health Organization (WHO) stated that "the frequency of bullying was estimated to be 8- 30 % and may reach 50% in many studies and In Egypt, the prevalence of bullying according to UNICEF was 77.8% among adolescent rural school students in other words 1 in 3 students experience bullying regularly, a recent study in Egypt showed the prevalence of bullying and victimization was high (67.5%) among studied group.

Deleterious oral habits are one of the public health problems that are commonly seen among children, it is defined as repeated orofacial muscular activities without a functional benefit Deleterious oral habits depend mainly on frequency, onset, and duration of habit which causes malocclusion such as open bite, deep bite, crossbite, and overjet that affects children's quality of life and cause psychological and esthetic problem, recent study In Alexandria, Egypt found that most seen oral habits in age 6 to 12 years are nail-biting 41.07% then tongue thrust 29.4% then mouth breathing with 15.9% and the least thumb sucking with 15.1%.

Children exposed to emotional stress and anxiety as bullying or need for comfort is considered as a main contributing factor to having an oral habit as children use oral habit as a source of safety and as a mechanism to release tension, pain, and anger through it. It is seen in children as bruxism, pacifier sucking, thumb sucking, mouth breathing, tongue thrusting, lip sucking, and biting and nail-biting.

Children at age of 8 years start to interact more with each other and become more observed so dental appearance becomes a site for bullying. the relationship between oral habit and bullying should be investigated because this type of abuse is a huge problem with serious psychosocial problems, Where the prevalence of children/adolescents being bullied ranges from 5.7% to 20.6%, bullied students are more likely to experience serious academic, social, psychological, and oral health problems there for more research into bullying is required to develop effective bullying prevention programs.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 8 to 10 years
2. Children who attended schools
3. Egyptian children

Exclusion Criteria:

1. Children who were taking antidepressants and anticonvulsant drugs
2. Children with cognitive/neurological disorders
3. Children with any syndromes such as ectodermal dysplasia or Down syndrome
4. Children with a history of an obvious alternative cause for malocclusion (e.g., trauma)
5. Participants' caregivers refuse to give consent

Ages: 8 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Egyptian school children, aged between 8-10 years, who attend school and their parents
Sampling Method: Non-Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Presence, duration, and frequency of Oral habits (Bruxism, Nail biting) | baseline
  Measure presence, duration, and frequency of Oral habits (Bruxism, Nail biting) through a questionnaire answered by parent including 3 questions with answeres yes and no or a. Did not notice in the past couple of months b. Only once or twice c. 2 or 3 times a month d. About once a week e. Several times a week

SECONDARY OUTCOMES:
Prevalence of Bullying and victimization | baseline
  Measure Prevalence of Bullying and victimization through a questionnaire answered by the child

REFERENCES:
- [Background] Weng X, Chui WH, Liu L. Bullying Behaviors among Macanese Adolescents-Association with Psychosocial Variables. Int J Environ Res Public Health. 2017 Aug 7;14(8):887. doi: 10.3390/ijerph14080887. PMID 28783110
- [Background] Alonso LS, Serra-Negra JM, Abreu LG, Martins IM, Tourino LFPG, Vale MP. Association between possible awake bruxism and bullying among 8- to 11-year-old children/adolescents. Int J Paediatr Dent. 2022 Jan;32(1):41-48. doi: 10.1111/ipd.12789. Epub 2021 May 7. PMID 33730369
- [Background] Ahmed GK, Metwaly NA, Elbeh K, Galal MS, Shaaban I. Prevalence of school bullying and its relationship with attention deficit-hyperactivity disorder and conduct disorder: a cross-sectional study. Egypt J Neurol Psychiatr Neurosurg. 2022;58(1):60. doi: 10.1186/s41983-022-00494-6. Epub 2022 May 23. PMID 35645553
- [Background] Kyriakides L, Kaloyirou C, Lindsay G. An analysis of the Revised Olweus Bully/Victim Questionnaire using the Rasch measurement model. Br J Educ Psychol. 2006 Dec;76(Pt 4):781-801. doi: 10.1348/000709905X53499. PMID 17094886
- [Background] Gaete J, Valenzuela D, Godoy MI, Rojas-Barahona CA, Salmivalli C, Araya R. Validation of the Revised Olweus Bully/Victim Questionnaire (OBVQ-R) Among Adolescents in Chile. Front Psychol. 2021 Apr 12;12:578661. doi: 10.3389/fpsyg.2021.578661. eCollection 2021. PMID 33912096
- [Background] Beckman L, Hellstrom L, von Kobyletzki L. Cyber bullying among children with neurodevelopmental disorders: A systematic review. Scand J Psychol. 2020 Feb;61(1):54-67. doi: 10.1111/sjop.12525. Epub 2019 Feb 28. PMID 30820957
- [Background] Dubey VP, Kievisiene J, Rauckiene-Michealsson A, Norkiene S, Razbadauskas A, Agostinis-Sobrinho C. Bullying and Health Related Quality of Life among Adolescents-A Systematic Review. Children (Basel). 2022 May 24;9(6):766. doi: 10.3390/children9060766. PMID 35740703
- [Background] Gomez-Baya D, Garcia-Moro FJ, Nicoletti JA, Lago-Urbano R. A Cross-National Analysis of the Effects by Bullying and School Exclusion on Subjective Happiness in 10-Year-Old Children. Children (Basel). 2022 Feb 18;9(2):287. doi: 10.3390/children9020287. PMID 35205007
- [Background] Lobbezoo F, Ahlberg J, Raphael KG, Wetselaar P, Glaros AG, Kato T, Santiago V, Winocur E, De Laat A, De Leeuw R, Koyano K, Lavigne GJ, Svensson P, Manfredini D. International consensus on the assessment of bruxism: Report of a work in progress. J Oral Rehabil. 2018 Nov;45(11):837-844. doi: 10.1111/joor.12663. Epub 2018 Jun 21. PMID 29926505
- [Background] Stewart RW, Drescher CF, Maack DJ, Ebesutani C, Young J. The Development and Psychometric Investigation of the Cyberbullying Scale. J Interpers Violence. 2014 Aug;29(12):2218-2238. doi: 10.1177/0886260513517552. Epub 2014 Jan 14. PMID 24424252
- [Background] Hayat MJ, Powell A, Johnson T, Cadwell BL. Statistical methods used in the public health literature and implications for training of public health professionals. PLoS One. 2017 Jun 7;12(6):e0179032. doi: 10.1371/journal.pone.0179032. eCollection 2017. PMID 28591190
- See also: School violence and bullying: Global status and trends, drivers and consequences — http://www.infocoponline.es/pdf/BULLYING.pdf
- See also: New UNESCO Report on School Violence and Bullying to be released at International Symposium on issue affecting millions worldwide — https://en.unesco.org/news/new-unesco-report-school-violence-and-bullying-be-released-international-symposium-issue
- See also: VIOLENCE AGAINST CHILDREN IN EGYPT Quantitative Survey and Qualitative Study in Cairo, Alexandria and Assiut — https://www.unicef.org/egypt/media/1906/file/Violence%20Against%20Children%20in%20Egypt-EN.pdf
- See also: Bullying and Victimization among Adolescents in Governmental Schools in Aswan City, Upper Egypt — https://ejcm.journals.ekb.eg/article_202266_bd56df488f1321d588779a69ba4143a4.pdf
- See also: Prevalence of oral habits among a group of Egyptian school children, and their knowledge regarding its bad effect on oral health — https://journals.ekb.eg/article_96994_42c3b3328b428c5e1f2d83df99608a1e.pdf
- See also: PREVELANCE OF DIFFERENT TYPES OF ORAL HABITS AMONG SCHOOL-CHILDREN AGED 6-12 YEARS IN ALEXANDRIA (A SURVEY STUDY) — https://eos.journals.ekb.eg/article_149880_c52a6066fe31ba0affd698f2ae6b2274.pdf
- See also: Deleterious Oral Habits among School Going Children - A Cross-Sectional Study — https://medicopublication.com/index.php/ijfmt/article/view/13145